CLINICAL TRIAL: NCT05884983
Title: Screening Effect of Dual-energy CT Combined With Nasopharyngeal Endoscopy for Screening Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Mingfang Ji, Clinical Professor, Zhongshan People's Hospital, Guangdong, China
Other Study IDs: NPC-PRO-004
Record Dates: First submitted 2023-05-04; First posted 2023-06-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Screening; Nasopharyngeal Carcinoma; Dual-energy CT; Endoscopy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endoscopy; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening cohort: 30-69 years old healthy participants in Zhongshan
  Interventions: Procedure: participants will undergo dual-energy CT and endoscopy

INTERVENTIONS:
Procedure: participants will undergo dual-energy CT and endoscopy — Diagnostic Test: P85-Ab,EBNA1-IgA,and VCA-IgA. Detect P85-Ab, EBNA1-IgA, VCA-IgA for all participants and select serological high-risk participants DiagnosticTest: dual-energy CT, endoscopy and biopsy. serological high-risk participants will refer to dual-energy CT, endoscopy and biospy
  Other Names: Biological/Vaccine: Blood and saliva Collect blood and saliva samples from participants

SUMMARY:
All participants will be tested for EBV-related biomarkers, including EBNA1-IgA, VCA-IgA, and BNLF2b total antibody (P85-Ab), and participants with high serologic risk will be selected based on serologic test results, and dual-energy CT will be performed first for high-risk screening subjects, and dual-energy CT will be performed first for the high-risk group to record dual-energy CT examinations of those suspected of nasopharyngeal carcinoma, and then endoscopy was performed on the high-risk group to record those suspected of nasopharyngeal carcinoma under endoscopy, and finally biopsies were taken for positive lesion sites indicated by dual-energy CT and suspicious lesion sites found by endoscopy to clarify the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject residents in Zhongshan City
* Subject has no medical record of nasopharyngeal carcinoma
* Subject is able to comprehend, sign, and date the written informed consent document to participate in the study
* Subject has psychical condition and well consciousness, and also accept and cooperate with the follow-up of this study

Exclusion Criteria:

* Subject has heavy cardiovascular, liver or kidney disease
* Subject has contraindications to nasopharyngeal endoscopy
* Subject has contrast media allergy

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30-69 years old healthy residences in Zhongshan City
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of dual-energy CT and endoscopy in the diagnosis of nasopharyngeal carcinoma | 6 months
  To compare the sensitivity [actual number of nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy / (actual number of nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy + number of nasopharyngeal cancers in the non-nasopharyngeal cancer population considered by dual-energy CT or endoscopy)] and specificity [actual number of non-nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy / ( actual number of non-nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy + number of non-nasopharyngeal cancers in the nasopharyngeal cancer population considered by dual-energy CT or endoscopy)] of dual-energy CT and endoscopy in the diagnosis of nasopharyngeal carcinoma, and to determine which test is more accurate in detecting nasopharyngeal carcinoma from the population
Positive and negative predictive values of dual-energy CT and endoscopy in the diagnosis of nasopharyngeal carcinoma | 6 months
  To compare the positive predictive value [actual number of nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy / (actual number of nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy + number of non-nasopharyngeal cancers in the nasopharyngeal cancer population considered by dual-energy CT or endoscopy )] and negative predictive value [actual number of non-nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy / (actual number of non-nasopharyngeal cancers in the population considered by dual-energy CT or endoscopy + number of nasopharyngeal cancers in the non-nasopharyngeal cancer population considered by dual-energy CT or endoscopy)] of dual-energy CT and endoscopy in the diagnosis of nasopharyngeal carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan People's Hospital, Zhongshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No